CLINICAL TRIAL: NCT04369742
Title: Treating COVID-19 With Hydroxychloroquine: A Multicenter Randomized, Double-blind, Placebo-controlled Clinical Trial in Hospitalized Adults
Brief Title: Treating COVID-19 With Hydroxychloroquine (TEACH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decision
Sponsor: NYU Langone Health (Other)
Collaborators: State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-00463
Record Dates: First submitted 2020-04-25; First posted 2020-04-30 (Actual); Results first posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, Randomized
Who Masked: Participant, Care Provider
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydroxychloroquine (Experimental)
  Interventions: Drug: Hydroxychloroquine (HCQ)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo: Calcium citrate

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ) — HCQ 400mg (2 tab) by mouth BID (day 1), 200mg (1 tab) by mouth BID (days 2-5)
  Arms: Hydroxychloroquine
Drug: Placebo: Calcium citrate — Calcium citrate 2 tablets (400mg) BID on day 1, 1 tablet (200mg) on days 2-5
  Arms: Placebo

SUMMARY:
Treatments for COVID-19 are urgently needed. Hydroxychloroquine (HCQ) is an antimalarial and immunomodulatory agent being repurposed for COVID-19 therapy based off in vitro data suggesting a possible antiviral effect. However, HCQ's effect on COVID-19 in human infection remains unknown. To fill this knowledge gap, we will enroll 626 adult patients hospitalized with laboratory-confirmed COVID-19 and randomize them 1:1 to a five-day course of HCQ or placebo. Notable exclusion criteria include ICU admission or ventilation on enrollment, prior therapy with HCQ, and baseline prolonged qTC. Our primary endpoint is a severe disease progression composite outcome (death, ICU admission, mechanical ventilation, ECMO, , and/or vasopressor requirement) at the 14-day post-treatment evaluation. Notable secondary clinical outcomes include 30-day mortality, hospital length of stay, noninvasive ventilator support, and cytokine release syndrome (CRS) grading scale. Secondary exploratory objectives will examine SARS-CoV-2 viral eradication at the EOT, changes in COVID-19 putative prognostic markers and cytokine levels, and titers of anti-SARS-CoV-2 antibodies. This randomized trial will determine if HCQ is effective as treatment in hospitalized non-ICU patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Hospitalized adult (≥18 years old) with symptoms consistent with COVID-19 including but not limited to any of the following: fever (documented or subjective), cough, dyspnea, diarrhea, nausea, diffuse myalgias, and/or anosmia
2. Informed consent signed by patient
3. Positive SARS-CoV-2 RT-PCR testing (nasopharyngeal, oropharyngeal, sputum and/or bronchoalveolar lavage) o The testing may:

   * Occur up to ≤72h prior to informed consent of participation in the study
   * Be undertaken either on-site or in an external laboratory certified by New York State to run testing for SARS-CoV-2

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Presence of the primary endpoint (ICU admission, mechanical ventilation, ECMO, and/or vasopressor requirement) at time of randomization.
2. Treatment with CQ or HCQ within the 30 days prior to the start of the study drug treatment.
3. Participation in a clinical trial to investigate a non-FDA approved drug with the intent to treat SARS-CoV-2 within the 30 days prior to the start of the study drug treatment.
4. Unable to take oral medications.
5. History of allergic reaction or intolerance to CQ or HCQ.
6. Baseline corrected qT interval >470 milliseconds (male) or >480 milliseconds (female), history of congenital qT prolongation, and/or history of cardiac arrest.
7. Concomitant therapy with flecainide, amiodarone, digoxin, procainamide, propafenone, thioridazine, or pimozide
8. History of retinal disease including a documented history of diabetic retinopathy.
9. Known history of G6PD deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mulligan, MD, FIDSA, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - State University of New York (SUNY) Downstate Medical Center, Brooklyn, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [contact information for PI or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to mark.mulligan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo
Started | 67 | 61
Completed | 53 | 50
Not Completed | 14 | 11
Not completed — Lost to Follow-Up (Day 14) | 7 | 4
Not completed — Lost to Follow-Up (Day 30) | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo | Total
Number analyzed (Participants) | 67 | 61 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (16.4) | 65.8 (16) | 66.2 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 45 | 31 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 25 | 50
  Not Hispanic or Latino | 42 | 36 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 11 | 25
  White | 23 | 18 | 41
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With SAE Through Day 30
Description: The measure value is reported as a percentage (# of patients with outcome/ # of patients * 100)
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 67 | 61
percentage of participants | 14.90 | 16.40

2. Primary Outcome: Percent of Participants With Grade 3 or 4 AEs Through Day 30
Description: The measure value is reported as a percentage (# of patients with outcome/ # of patients * 100)
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 67 | 61
percentage of participants | 13.40 | 13.10

3. Primary Outcome: Percent of Participants With Discontinuation of Therapy (for Any Reason)
Description: The measure value is reported as a percentage (# of patients with outcome/ # of patients * 100)
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 67 | 61
percentage of participants | 23.90 | 24.6

4. Primary Outcome: Percent of Participants Showing a Severe Disease Progression Composite Outcome
Description: Including any of the following: mortality, ICU admission, invasive mechanical ventilation, ECMO, and/or hypotension requiring vasopressor support by the 14-day post-treatment evaluation (PTE). The measure value is reported as a percentage (# of patients with outcome/ # of patients * 100).
Time Frame: 14 days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 60 | 57
percentage of participants | 18.30 | 10.50

5. Secondary Outcome: Hospital Length of Stay
Description: LOS is defined as the interval (in days) that the patient was admitted to a non-rehabilitation floor, categorized as short (<7 days), moderate (7-10 days), or extended (>10 days)
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 67 | 61
days | 9.75 (10.3) | 6.8 (5.92)

6. Secondary Outcome: Days of Fever
Description: Defined as number of days with temperature >100.4 degrees Fahrenheit.
Time Frame: 14 days
Measure: Median (Full Range); unit: days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 67 | 59
days | 0 [0 to 5] | 0 [0 to 6]

7. Secondary Outcome: Days of Non-invasive Ventilator Use
Description: Defined as days the patient is placed on non-invasive ventilator support (CPAP or BiPAP), excluding routine CPAP use for sleep apnea.
Time Frame: 14 days
Measure: Median (Full Range); unit: days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 67 | 61
days | 0 [0 to 4] | 0 [0 to 1]

8. Secondary Outcome: Days of Non-rebreather Mask Oxygen Supplementation
Description: Defined as the number of days the subject was on a non-rebreather mask.
Time Frame: 14 days
Measure: Median (Full Range); unit: days
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 67 | 61
days | 0 [0 to 6] | 0 [0 to 7]

9. Secondary Outcome: Number of Participants With Mild, Moderate, and Severe Scores on Cytokine Release Syndrome (CRS) Grading Scale
Description: Grade 1 (mild) = able to be managed with nonparenteral supportive care, Grade 2 (moderate) = at least one of the following present (hospitalization needed for management of CRS-related symptoms, parenteral nutrition or supportive care required, signs of moderate/severe organ dysfunction), Grade 3 (severe) = hospitalization needed for management of at least one of the following (hypotension, hypoxia, organ dysfunction, coagulopathy), Grade 4 (life-threatening) = at least one of the following present (hypotension requiring high-dose vasopressors, hypoxia requiring mechanical ventilation).
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 67 | 61
Participants
  Mild | 27 | 21
  Moderate | 25 | 33
  Severe | 15 | 7

10. Secondary Outcome: Percent of Subjects With Q-T Interval, Corrected (qTC) Prolongation at End of Treatment (EOT)
Description: (≥470 milliseconds in men; ≥480 milliseconds in women) on electrocardiogram at EOT (Day 6)
Time Frame: 6 Days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 41 | 39
percentage of participants | 24.4 | 12.8

11. Secondary Outcome: Percent of Patients Who Resulted in Mortality
Description: Individual component of severe disease progression composite endpoint evaluated. The measure value is reported as a percentage (# of patients with outcome/ # of patients * 100).
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 53 | 50
percentage of participants | 13.2 | 12

12. Secondary Outcome: Percent of Participants Who Required ICU Admission
Description: as for outcome 11
Time Frame: 30 Days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 53 | 50
percentage of participants | 17 | 6

13. Secondary Outcome: Percent of Participants Who Required Invasive Mechanical Ventilation
Description: as for outcome 11
Time Frame: 30 Days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 53 | 50
percentage of participants | 9 | 6

14. Secondary Outcome: Percent of Participants Who Required Extracorporeal Membrane Oxygenation (ECMO)
Description: as for outcome 11
Time Frame: 30 Days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 53 | 50
percentage of participants | 0 | 0

15. Secondary Outcome: Percent of Participants With Hypotension Requiring Vasopressor Support
Description: Individual component of severe disease progression composite endpoint evaluated. For incidence, the measure value is reported as a percentage (# of patients with outcome/ # of patients * 100)
Time Frame: 30 Days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 53 | 50
percentage of participants | 3.77 | 4

16. Secondary Outcome: Percent of Participants With SARS-CoV-2 Viral Eradication From Nasopharyngeal Specimens at EOT
Description: Laboratory endpoint, measured by RT-PCR, reported as the percentage of negative results at day 6
Time Frame: 6 days
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 37 | 30
percentage of participants | 21.60 | 33.30

17. Secondary Outcome: Change in Alanine Aminotransferase (ALT) Levels
Description: Biochemistry lab-work will be completed to obtain ALT levels (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 58 | 44
U/L | 19.3 (52.8) | 8.3 (30.4)

18. Secondary Outcome: Change in Aspartate Aminotransferase (AST) Levels
Description: Biochemistry lab-work will be completed to obtain AST levels (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 58 | 44
U/L | -1.52 (66.2) | 3.66 (35.3)

19. Secondary Outcome: Change in Creatinine Levels
Description: Biochemistry lab-work will be completed to obtain Creatinine levels (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 64 | 57
mg/dL | 0.0198 (1.2) | -0.169 (1.19)

20. Secondary Outcome: Change in Glucose Levels
Description: Biochemistry lab-work will be completed to obtain Glucose levels (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 64 | 56
mg/dL | 2.69 (47.4) | -15.7 (39.7)

21. Secondary Outcome: Change in White Blood Cell (WBC) Count
Description: Hematology lab-work will be completed to obtain WBC count (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: cells per 10^6 L
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 63 | 56
cells per 10^6 L | -0.0868 (3.86) | -0.0839 (3.27)

22. Secondary Outcome: Change in Hemoglobin Levels
Description: Hematology lab-work will be completed to obtain hemoglobin levels (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: gm/dL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 63 | 56
gm/dL | -0.5 (1.07) | -0.443 (1.17)

23. Secondary Outcome: Change in Platelet Count
Description: Hematology lab-work will be completed to obtain platelet count (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: platelets per 10^6 L
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 63 | 56
platelets per 10^6 L | 63.4 (110) | 65.8 (100)

24. Secondary Outcome: Change in Total Bilirubin Levels
Description: Biochemistry lab-work will be completed to obtain bilirubin levels (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 52 | 43
mg/dL | -0.183 (0.819) | -0.0509 (0.619)

25. Secondary Outcome: Change in Lactate Dehydrogenase (LDH) Levels
Description: Biochemistry lab-work will be completed to obtain LDH levels (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 53 | 52
U/L | -2.65 (153) | -45.1 (162)

26. Secondary Outcome: Change in C-Reactive Protein (CRP) Levels
Description: Biochemistry lab-work will be completed to obtain CRP levels (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 55 | 50
mg/L | -21.8 (77.7) | -23.8 (113)

27. Secondary Outcome: Change in Interleukin 6 (IL-6) Levels
Description: Biochemistry lab-work will be completed to obtain IL-6 levels (if not obtained as part of routine clinical care, the research team will order for clinical lab to add onto remnant specimens, if available).
Time Frame: Baseline, 6 days
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 25 | 19
pg/ml | 85.6 (245) | 19.3 (101)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Regular investigator assessment (monitoring for unsolicited adverse events days 1-5, recording of solicited adverse events at days 6, 14, and 30)
Arm/Group | Hydroxychloroquine | Placebo
All-Cause Mortality (participants affected / at risk) | 7/67 | 6/61
Serious Adverse Events (participants affected / at risk) | 10/67 | 10/61
Other Adverse Events (participants affected / at risk) | 32/67 | 30/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydroxychloroquine (N=67) | Placebo (N=61)
Acute renal failure (Renal and urinary disorders) | 1 | 1
Alcohol withdrawal syndrome (General disorders) | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 1 | 0
Congestive heart failure (Cardiac disorders) | 1 | 0
Death (General disorders) | 7 | 6
Diverticulitis (Infections and infestations) | 0 | 1
Electrocardiogram QTc interval prolonged (Cardiac disorders) | 1 | 0
Hospice care (General disorders) | 0 | 1
Hospital acquired hyponatremia (Infections and infestations) | 1 | 0
Hospitalization (General disorders) | 0 | 1
Hyperkalemia (General disorders) | 0 | 1
Intra-abdominal abscess (Infections and infestations) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolus (Blood and lymphatic system disorders) | 0 | 1
stroke (Nervous system disorders) | 1 | 0
Subdural hematoma (Nervous system disorders) | 1 | 0
Subdural hemorrhage (Nervous system disorders) | 1 | 0
Syncope (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydroxychloroquine (N=67) | Placebo (N=61)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 2
Bleeding vaginal (Reproductive system and breast disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 4
Deliria (incl confusion) (General disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Diabetes mellitus (incl subtypes) (Endocrine disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 4
Dry mouth (Skin and subcutaneous tissue disorders) | 1 | 0
DVT (Blood and lymphatic system disorders) | 0 | 1
Electrocardiogram QTc interval prolonged (Cardiac disorders) | 2 | 1
Electrolytes NOS abnormal (General disorders) | 1 | 1
Elevated liver enzyme levels (Hepatobiliary disorders) | 1 | 0
Epistaxis (General disorders) | 0 | 1
Fall (General disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Hematoma (General disorders) | 0 | 1
Hives (Immune system disorders) | 0 | 1
Hyperkalemia (General disorders) | 0 | 3
Hypokalemia (General disorders) | 2 | 2
Hypomagnesemia (General disorders) | 1 | 0
Hyponatremia (General disorders) | 0 | 1
Hypotension (General disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Injection site pain (Skin and subcutaneous tissue disorders) | 0 | 1
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea and/or vomiting (Gastrointestinal disorders) | 7 | 2
Non-sustained ventricular tachycardia (Cardiac disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Staphylococcal pneumonia (Infections and infestations) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Syncope (General disorders) | 1 | 0
Vaginal yeast infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04369742/Prot_SAP_000.pdf